CLINICAL TRIAL: NCT04470674
Title: Randomized Phase II Study of Durvalumab or Durvalumab Plus Chemotherapy in Kras Mutation Positive and PD-L1 High (≥ 50%) NSCLC Patients
Brief Title: Study of Durvalumab or Durvalumab Plus Chemotherapy in Kras Mutation Positive and PD-L1 High (≥ 50%) NSCLC Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Accrual
Sponsor: Shirish M Gadgeel (Other)
Collaborators: AstraZeneca (Industry); Henry Ford Health System (Other)
Responsible Party: Sponsor-Investigator, Shirish M Gadgeel, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCRN LUN17-126
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Lung Cancer; Non-small Cell Lung Cancer; PD-L1 Gene Mutation; KRAS Activating Mutation
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (Durvalumab) (Active Comparator): Durvalumab 1500 mg IV every 4 weeks for 13 cycles.
  Interventions: Drug: Durvalumab
- Arm B (Durvalumab plus chemotherapy) (Experimental): Durvalumab 1500 mg IV plus carboplatin AUC 5 IV and pemetrexed 500 mg/m2 IV every 3 weeks for 4 cycles followed by durvalumab and pemetrexed every 3 weeks for 13 more cycles.
  Interventions: Drug: Durvalumab; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500 mg
  Other Names: IMFINZI
Drug: Carboplatin — carboplatin AUC 5
  Arms: Arm B (Durvalumab plus chemotherapy)
Drug: Pemetrexed — pemetrexed 500 mg/m2
  Other Names: Alimta
  Arms: Arm B (Durvalumab plus chemotherapy)

SUMMARY:
This is a two arm, randomized, phase II study of patients with advanced KRAS mutation positive and PD-L1 high NSCLC who have not received therapy for advanced stage disease. Patients will be randomized between Arm A and Arm B treatment. Arm A treatment will consist of durvalumab every 4 weeks for 13 cycles. Arm B treatment will consist of durvalumab with chemotherapy every 3 weeks for 4 cycles followed by durvalumab with pemetrexed every 3 weeks for 13 cycles.

ELIGIBILITY:
Inclusion Criteria

* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* Body weight > 30 kg. If body weight falls to 30 kg or below during the study, the subject will be removed from study drugs.
* ECOG Performance Status of 0-1 within 7 days prior to registration.
* Life expectancy of ≥ 12 weeks.
* Histological or cytological evidence of stage IV Kras mutation positive non-squamous NSCLC.
* Patients who have recurrence following treatment for earlier stages of NSCLC are eligible provided the recurrence has not occurred within 12 months of completing prior therapy.
* Patient's tumor must be known to be PD-L1 high (≥ 50%). SP-142 assay will not be accepted. See Section 8.1 for additional information regarding this result.
* Measurable disease according to RECIST v1.1 criteria within 4 weeks of study registration.
* Demonstrate adequate organ function as defined in the table below; all screening labs to be obtained within 14 days prior to registration.

  * Absolute Neutrophil Count (ANC) ≥ 1.5 K/mm3
  * Hemoglobin (Hgb) ≥ 9.0 g/dL
  * Platelets ≥ 75 k/mm3
  * Calculated creatinine clearance ≥ 45 cc/min using the Cockcroft-Gault formula
  * Bilirubin ≤ 1.5 × upper limit of normal (ULN) This will not apply to subjects with clinical diagnosis of Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology)
  * Aspartate aminotransferase (AST) ≤ 2.5 × ULN, unless patients has liver metastases in which case it must be ≤5 × ULN
  * Alanine aminotransferase (ALT) ≤ 2.5 × ULN, unless patients has liver metastases in which case it must be ≤5 × ULN
* Evidence of post-menopausal status or negative urine or serum pregnancy test for female pre-menopausal patients. NOTE: Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. See section 5.4 for age-specific requirements (<50 year old vs. ≥50 year old).
* Females of childbearing potential randomized to Arm A and males randomized to Arm A or Arm B must be willing to abstain from heterosexual activity or agree to use a highly effective method of contraception from the time of informed consent until 90 days after treatment discontinuation. Females of childbearing potential randomized to Arm B must be willing to abstain from heterosexual activity or agree to use a highly effective method of contraception until 180 days after treatment discontinuation. See section 5.4 for definition of childbearing potential.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study

Exclusion Criteria

* Patient must not have received any prior systemic therapy for stage IV NSCLC. Patients must not have received prior anti-PD-1 or anti-PD-L1.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Testing is not required at screening.
* Patients with history of non-infectious pneumonitis that required steroids or has current pneumonitis. Has known history of Interstitial Lung Disease (ILD) or radiation pneumonitis which required therapy with steroids.
* Active or prior documented autoimmune or inflammatory (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis, systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]) and pneumonitis. The following are exceptions to this criterion:

  * Diverticulosis
  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study sponsor investigator.
  * Patients with celiac disease controlled by diet alone
* History of allogenic progenitor/stem cell or organ transplantation.
* History of immunodeficiency. Patient should not be on any immunosuppressive therapy or steroids > prednisone 10mg/day or its equivalent on the day of the start of therapy.
* Patients with current or prior use of immune suppressive therapy within 7 days of starting study therapy. Following exceptions are allowed

  * Intranasal, local (eg. Intraarticular injections), inhaled or topical steroids
  * Steroids to prevent hypersensitivity reactions, eg. IV contrast for CT scans
  * Systemic steroids not to exceed 10mg of prednisone or its equivalent.
* Any concurrent chemotherapy, investigational product, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* Patients who have received live attenuated vaccine within 30 days of the first dose of study therapy. Patients should not receive live vaccines while on therapy and for 30 days after the last dose.
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* History of another primary malignancy except for

  * Malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of IP and of low potential risk for recurrence. Patients with elevated PSA (prostate specific antigen) as the only evidence of prostate cancer may be considered for enrolment after discussion with the sponsor-investigator.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* Patients with leptomeningeal carcinomatosis are not eligible. Patients with symptomatic brain metastases are eligible only after receiving appropriate therapy, are clinically stable and do not require steroids equivalent to 10 mg of prednisone daily. Patients with asymptomatic brain metastases are eligible if the treating physician determines that the brain metastases do not require immediate directed therapy, they are clinically stable, and are not using steroids equivalent to >10mg of prednisone day prior to trial treatment.
* Any unresolved toxicity from previous anticancer therapy Grade ≥2 except for alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

  * Patients with Grade ≥ 2 neuropathy will be evaluated on a case-by-case basis after consultation with the sponsor-investigator.
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the sponsor-investigator.
* Patients who have radiation therapy within 1 week prior to Day 1. Patients should have recovered from any adverse events related to radiation therapy to ≤ grade 1 or baseline. Patients must be considered stable to receive study therapy.
* Participation in another clinical study with an investigational product within 30 days prior to study registration.
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* Major surgery as determined by the treating physician within 4 weeks of study registration. Placement of a central access device (port) is not considered major surgery.
* Uncontrolled intercurrent illness as determined by the treating physician, including but not limited to, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* History or hypersensitivity reaction to carboplatin, cisplatin or other platinum-containing compounds, pemetrexed, or durvalumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
Response Rate | 12 months
  Assess response rate by RECIST criteria 1.1 in Arm A and Arm B in advanced Kras mutation positive and PD-L1 high (≥50%) NSCLC patients.The objective response rate is the proportion of all subjects with confirmed PR or CR according to RECIST 1.1, from the start of treatment until disease progression/recurrence

SECONDARY OUTCOMES:
Progression Free Survival | 12 months
  A measurement from the date of randomization until the criteria for disease progression is met as defined by RECIST 1.1 or death occurs.
Assess adverse events | 12 months
  Adverse events will be summarized by frequency and severity using CTCAE version 5.
Overall Survival | 12 months
  Overall survival is defined by the date of randomization to date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Shirish M Gadgeel, MBBS, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No